CLINICAL TRIAL: NCT02976298
Title: Rôle du Cervelet et de l'Aire Motrice supplémentaire Dans le contrôle Postural au Cours de la Marche Chez l'Homme
Brief Title: Effects of Cerebellum or Supplementary Motor Area Functional Inactivation on Gait and Balance Control
Acronym: CERESMARCHE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C12-05; 2012-A00796-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-03-26; First posted 2016-11-29 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2016-11

CONDITIONS: Transcranial Magnetic Stimulation
Keywords: cerebellum; supplementary motor area
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- transcranial magnetic stimulation (Sham Comparator): sham transcranial magnetic stimulation
  Interventions: Other: transcranial magnetic stimulation
- supplementary motor area stimulation (Experimental): supplementary motor area transcranial magnetic stimulation
  Interventions: Other: transcranial magnetic stimulation
- cerebellar stimulation (Experimental): cerebellar transcranial magnetic stimulation
  Interventions: Other: transcranial magnetic stimulation

INTERVENTIONS:
Other: transcranial magnetic stimulation — comparison of different conditions of transcranial magnetic stimulation

SUMMARY:
In human, the physiology of gait and balance is not clearly established. By using functional imaging and electrophysiological techniques, various brain regions from the cortex to the midbrain area, including the cerebellum, have been identified as involved in such control. The specific role of these structures in both the capacity to go forward (locomotion) and stand upright (balance), but also in the different phases of the gait initiation process, are not known, however. In this study,the investigators aimed to assess the specific role of both the supplementary motor area (SMA) and the cerebellum in postural control during the initiation of gait. For this purpose, the investigators plan to study the gait initiation in 20 healthy subjects before and after functional inactivation (using inhibitory repetitive transcranial magnetic stimulation, rTMS) of the cerebellum or SMA. Biomechanical, kinematic and electromyographic parameters of the gait initiation will be recorded using a force platform, reflective markers with infrared cameras (VICON system) and lower limbs surface EMG electrodes.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* agree to participate to the study with signature of the informed consent
* heathy insurance
* normal clinical exam

Exclusion Criteria:

* previous medical history of neurological, rheumatological, orthopedic or psychiatric disorders
* contra-indication to MRI or TMS
* drug treatment that modifies the nervous central system excitability (antidepressant, antiepileptic, neuroleptic)
* chronic alcoholism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
postural control during gait initiation | change between baseline and 5 minutes after transcranial magnetic stimulation
  braking capacity

SECONDARY OUTCOMES:
duration of anticipatory postural adjustments | change between baseline and 5 minutes after transcranial magnetic stimulation
  duration

OTHER OUTCOMES:
centre of foot pressure displacement during postural adjustments | change between baseline and 5 minutes after transcranial magnetic stimulation
  centre of foot pressure displacement measured by force platform
step length | change between baseline and 5 minutes after transcranial magnetic stimulation
  step length
step velocity | change between baseline and 5 minutes after transcranial magnetic stimulation
  step velocity
duration of electromyographic activity of the tibialis anterior muscles | change between baseline and 5 minutes after magnetic transcranial stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Welter, MD, PhD, Principal Investigator — APHP; Sabine Meunier, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- M.L.Welter, Paris, France

REFERENCES:
- [Background] Richard A, Van Hamme A, Drevelle X, Golmard JL, Meunier S, Welter ML. Contribution of the supplementary motor area and the cerebellum to the anticipatory postural adjustments and execution phases of human gait initiation. Neuroscience. 2017 Sep 1;358:181-189. doi: 10.1016/j.neuroscience.2017.06.047. Epub 2017 Jul 1. PMID 28673716